CLINICAL TRIAL: NCT00729222
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study of the Hemodynamic Effects of Rolofylline Injectable Emulsion in the Treatment of Patients With Heart Failure
Brief Title: Hemodynamic Effects of Rolofylline in the Treatment of Patients With Heart Failure (7418-503)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: NovaCardia, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7418-503; MK7418-503; 2008_532
Record Dates: First submitted 2008-08-05; First posted 2008-08-07 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — rolofylline

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: Placebo
- 2 (Experimental): rolofylline
  Interventions: Drug: rolofylline

INTERVENTIONS:
Drug: Comparator: Placebo — rolofylline placebo IV infusion over 4 hours.
  Arms: 1
Drug: rolofylline — rolofylline 30 mg IV infusion over 4 hours.
  Arms: 2

SUMMARY:
The study will estimate the effects of rolofylline, alone and in addition to loop diuretic therapy on pulmonary capillary wedge pressure and other hemodynamic parameters, in patients with heart failure and renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with heart failure and renal impairment, currently using furosemide, with systolic blood pressure >95 mm Hg

Exclusion Criteria:

* Patient has active infection, use of diuretic within 3 hours of screening visit, has acute tubular necrosis or severe pulmonary disease, any heart problems within the last two weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
change in pulmonary capillary wedge pressure | from baseline to 4 and 8 hours

SECONDARY OUTCOMES:
Change in cardiac output, systemic vascular resistance, pulmonary vascular resistance, pulmonary pressure and right atrial pressure | from baseline to 4 and 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Ponikowski P, Mitrovic V, O'Connor CM, Dittrich H, Cotter G, Massie BM, Givertz MM, Chen E, Murray M, Weatherley BD, Fujita KP, Metra M. Haemodynamic effects of rolofylline in the treatment of patients with heart failure and impaired renal function. Eur J Heart Fail. 2010 Nov;12(11):1238-46. doi: 10.1093/eurjhf/hfq137. Epub 2010 Sep 7. PMID 20823097